CLINICAL TRIAL: NCT05149170
Title: Radiotherapy With Inductive and Concurrent Anti-PD-1 Antibody in Early-stage Low-risk Extranodal NK/T Cell Lymphoma, Nasal Type: A Multi-center Phase II Study
Brief Title: Radiotherapy and Anti-PD-1 in Low-risk ES-ENKTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); The First Hospital of Jilin University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Shunan Qi, Associated Prof. in the radiation oncology department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCG-NKT-2101
Record Dates: First submitted 2021-11-06; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Early-stage; Extranodal NK-T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: NK/T-Cell Lymphoma, Nasal and Nasal-Type; radiotherapy; Anti-PD-1 Antibody
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — spartalizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inductive and concurrent anti-PD-1 antibody combined with radiotherapy (Experimental): All the enrolled patients receive 2 doses of inductive anti-PD-1 antibody (Tislelizumab 200mg) every two weeks, and then Involved-site radiotherapy (50±6-10 Gy) with concurrent anti-PD-1 antibody (Tislelizumab 200mg) every two weeks.
  Interventions: Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — inductive Anti-PD-1 antibody + concurrent Anti-PD-1 antibody with RT
  Other Names: radiotherapy

SUMMARY:
The current study is a phase II multi-center single arm trial to evaluate the efficacy and safety of adding Anti-PD-1 antibody in an inductive and concurrent way to radiotherapy in early-stage low-risk extranodal NK/T cell lymphoma, nasal type

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proved extranodal NK/T cell lymphoma
* No previous anti-cancer treatment
* Measurable lesion on baseline PET/CT and MRI
* Stage I
* Normal serum LDH level
* Primary tumor invasion (PTI) absence
* ECOG PS 0-1
* Sufficient organ functions

Exclusion Criteria:

* Other mature T- or NK- lymphoma
* Hemophagocytic lymphohistiocytosis
* Primary CNS lymphoma or CNS-involved lymphoma
* History of malignancy except for cutaneous basal-/squamous- cell carcinoma or cervical carcinoma in situ 3 years prior to study treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete response after inductive therapy | 2-4 weeks after inductive anti-PD-1 antibody
  complete resolution of disease in imaging and biopsy after inductive therapy

SECONDARY OUTCOMES:
Progression-free survival rate at year 2 after enrollment, 2y-PFS | 2-year
  From enrollment to any disease progression or death
Overall Survival rate at year 2/5 after enrollment，2y-/5y-OS | 2-year, 5-year
  From enrollment to death
Rate of acute toxicity (any and above grade 3) | From enrollment to 3 months after treatment
  toxicities according to CTCAE criteria
Quality of Life change, QoL | baseline, 1/3/6/12/24 months after treatment
  measurement basing on EORTC-QLQ-HN35 tables
Quality of Life change, QoL | baseline, 1/3/6/12/24 months after treatment
  measurement basing on EORTC-QLQ-C30 tables

OTHER OUTCOMES:
Biomarkers to predict anti-PD-1 antibody efficacy and 2y-PFS | baseline
  potential biomarkers in baseline tumor samples and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Ye-Xiong Li, MD, Principal Investigator — CAMS
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From: 6 months after publication. To: 5 years after publication
Access Criteria: Will share data with the PIs who had specific study plan in immunotherapy area and biomarker area

REFERENCES:
- [Derived] Li JY, Qi SN, Hu C, Liu X, Yang Y, Wu T, Zheng R, Feng XL, Ni XG, Jin FY, Song YQ, Liu WP, Zhou SY, Li YX. Tislelizumab and radiation therapy in low-risk early-stage extranodal natural killer/T-cell lymphoma, nasal type: a phase II study protocol. Future Oncol. 2024 Feb;20(5):245-256. doi: 10.2217/fon-2023-0065. Epub 2023 Nov 29. PMID 38018460